CLINICAL TRIAL: NCT01054794
Title: Temporary Gastric Neurostimulation for Gastroparesis
Brief Title: Temporary Gastric Electrical Stimulation for Gastroparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Christopher Andrews, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TS01
Record Dates: First submitted 2010-01-19; First posted 2010-01-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Gastric Electrical Stimulation
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation ON (Active Comparator)
  Interventions: Device: Gastric mucosal stimulation
- Stimulation OFF (Sham Comparator)
  Interventions: Device: Gastric mucosal stimulation

INTERVENTIONS:
Device: Gastric mucosal stimulation — The lead is a sterile, 2mm diameter insulated wire (Temporary Transvenous Pacing Lead 6416-200cm, Medtronic, Minneapolis, MN) with 2 electrodes on the distal end. The mucosal stimulation parameters(Current:10 mA; Frequency: 14Hz; Pulse width: 330 ms; Cycle ON: 0.1 s; Cycle OFF: 5 s) are within the range used for standard permanent implanted GES (Enterra therapy) within the serosa and muscle layers of the stomach, and which has been shown to be safe, without any tissue damage.

SUMMARY:
This is a prospective study of temporary gastric mucosal electrical stimulation (tGES) in 30 patients with gastroparesis (GP). After a 7 day baseline assessment of symptoms, subjects will have an endoscopically-placed tGES lead implanted into the mucosa of the antrum. This lead is connected to a thin wire that runs up the esophagus and out the nostril, similar to a nasojejunal feeding tube, although much thinner. It is then attached to a programmable battery pack which provides the desired level of stimulation.

Patients will then be randomized to 7 days OFF or 7 days ON stimulation in a double-blind fashion. After 7 days, subjects will crossover to the other study arm (ie ON patients will be switched off; OFF patients will be switched on). Symptoms and QoL measures will be assessed at baseline, ON, and OFF periods. Serum ghrelin and other hormones, as well as EGG will be assayed after 6 days in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older
* Existing clinical diagnosis of gastroparesis for at least one year as judged by the study gastroenterologist based on past medical history, clinical symptoms
* Sufficiently symptomatic at time of proposed study (Minimum total baseline GCSI score of 1.5 or higher)
* Delayed gastric emptying (>10% retention at 4 hours) on standard scintigraphic emptying study with patients off narcotics for at least 48 hours. Normal upper endoscopy (with the exception of small bezoars) since the onset of symptoms
* Medically fit to undergo endoscopy
* Able and willing to remain in Calgary for the duration of the study (baseline period excepted)
* Able to provide written informed consent

Exclusion Criteria:

* Clinical evidence (including physical exam and/or EKG) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns
* Current use of anticoagulants, ASA, NSAIDS, clopidogrel, etc. which cannot safely be stopped for up to 5 days prior to the procedure in the opinion of the investigators
* Bleeding diathesis
* Severe immunocompromise
* Physical, mental, or compliance issues which in the opinion of the investigators may prevent the patient from completing the study
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in patient symptoms during the ON and OFF periods of tGES stimulation. | daily x 6 days in each phase of study (ON and OFF)

SECONDARY OUTCOMES:
1. Changes in serum ghrelin and leptin between ON and OFF periods of tGES stimulation in GP patients. 2. Changes in gastric electrical activity between ON and OFF periods of tGES stimulation in GP patients | Once during each study phase (ON and OFF)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Andrews, MD, FRCPC, Principal Investigator — University of Calgary, Faculty of Medicine
Locations (1):
- University of Calgary, Calgary, Alberta, Canada